CLINICAL TRIAL: NCT07139483
Title: Preventing Chronification of Phantom Limb Pain Through Mirror Therapy in Conjunction With Transcranial Direct Current Stimulation
Brief Title: Preventing Chronification of Phantom Limb Pain Through Mirror Therapy in Conjunction With tDCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Collaborators: Loewenstein Hospital (Other); Reuth Rehabilitation Hospital (Other); Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 253/23
Record Dates: First submitted 2025-05-21; First posted 2025-08-24 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Phantom Limb Pain After Amputation
Keywords: PLP; Phantom sensation; telescoping; amputation; tDCS; MT; Maladaptive plasticity; Phantom Limb Pain
MeSH Terms: conditions — Phantom Limb | interventions — Mirror Movement Therapy

STUDY DESIGN:
Intervention Model Description: The study consists of 2 main parallel participants groups: traumatic and a-traumatic. Upon their arrival at the rehabilitation centers, participants will be recruited, give consent, and receive a serial number. Only patients developing PLP will be randomly assigned to the study arms.
  There will be 3 randomized patient arms (for each participants group): (1) no-intervention, natural-course group; (2) MT + sham tDCS; (3) MT + real tDCS . Therefore, the proposed project is a randomized, controlled, double blind, multicenter study. Further, the personnel collecting the data will be fully blinded to group assignments.
  The data will be collected at 5 timepoints during the experiment. Each timepoint will comprise 1 week of assessments: T1 (baseline week), before the 4 weeks of neuromodulatory application; T2, immediately after the end of the application; and T3, T4, and T5, assessments conducted 1, 3, and 6 months, respectively, after the end of the neuromodulatory application
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mirror Therapy + real tDCS (Active Comparator): Both MT and tDCS neuromodulatory interferences (separately or combined) will consist of 20 sessions, each lasting 20 min, completed during 4 weeks, once daily (excluding weekends). The neuromodulatory interferences will be self-administered by the participants. The first 2 sessions (at the clinic) will include training to familiarize participants (and their primary caregivers) with the procedure and to instruct them on the self-administering techniques that the researchers and others successfully employed. After training, neuromodulatory interferences will be applied either at the clinic (during hospitalization) or at home (after discharge). This approach promotes participants' retention and reduces dropouts, especially when the study constitutes multiple sessions.
  Interventions: Device: Trans Direct-Cranial Stimulation (tDCS); Behavioral: Mirror therapy
- Mirror Therapy + sham tDCS (Sham Comparator): Both MT and tDCS neuromodulatory interferences (separately or combined) will consist of 20 sessions, each lasting 20 min, completed during 4 weeks, once daily (excluding weekends). The sham tDCS will be identical to the real tDCS, except no current will be applied. However, as recommended, during the first and last 30 sec, the current will be ramped up to 1.5 mA and immediately back to 0 to induce scalp sensations similar to those in real tDCS, further supporting blinding
  Interventions: Device: Trans Direct-Cranial Stimulation (tDCS); Behavioral: Mirror therapy
- No-intervention, natural-course group (No Intervention): The participants will receive the regular treatment regimen at the rehabilitation center, including physical-therapy and pharmacological treatment, without intervention of Mirror-therapy and tDCS.

INTERVENTIONS:
Device: Trans Direct-Cranial Stimulation (tDCS) — The tDCS electrodes will be inserted into 5×7 cm (35 cm2) sponges soaked with saline (0.9 M) and placed as follows: anode over the M1 contralateral to the amputated limb (adjusted based on lower/upper amputation), and cathode over the forehead, contralateral to the anode (ipsilateral to amputated limb). Total stimulation duration will be 20 min, with a rise and decline time of 30 sec and stimulus intensity of 1.5 mA for the real tDCS real. The intensity of 1.5 mA is in the midrange of recommended intensities (1-2 mA) and supports successful blinding. The sham tDCS will be identical to the real tDCS, except no current will be applied. However, as recommended, during the first and last 30 sec, the current will be ramped up to 1.5 mA and immediately back to 0 to induce scalp sensations similar to those in real tDCS, further supporting blinding. The Mini-CT tDCS Stimulator device has been developed for home use and allows double-blind administration.
  Arms: Mirror Therapy + real tDCS; Mirror Therapy + sham tDCS
Behavioral: Mirror therapy — Participants will be seated with a portable mirror between their limbs so that the unaffected limb is reflected in the mirror. The participants will focus their attention on the reflection in the mirror and perform the following movements: plantarflexion and dorsiflexion and inversion and eversion of the foot, flexion and extension of the wrist and ulnar and radial deviation, for lower and upper limp amputates, respectively. The participants will continue performing the 2 sets of movements for 20 minutes (with short intermissions if needed)
  Arms: Mirror Therapy + real tDCS; Mirror Therapy + sham tDCS

SUMMARY:
Background: Most amputees experience phantom limb pain (PLP), for years after amputation. Virtually all PLP research to date has focused on the mechanisms of chronic PLP, ignoring the mechanisms of chronification. This research project will focus on combined neuromodulatory interventions of mirror therapy (MT) and trans direct-cranial stimulation (tDCS), applied for the first time at the acute state of PLP, with an aim to prevent its chronification and chronicity. In PLP, maladaptive plasticity associated with sensory deafferentation following an amputation is one of the contributors for excessive pain.

MT is a well-accepted yet limited option, which is thought to counterbalance abnormal plasticity. tDCS is an emerging approach believed to affect the membrane potential and activity threshold of cortical neurons. tDCS analgesic effectiveness, however, is mild and short, rendering it a noneffective stand-alone treatment. The researchers' objectives are to investigate whether the combined therapy of MT and tDCS will prevent chronic PLP and improve its related clinical characteristics. In addition, the researchers will investigate the behavioral manifestations effects of the combined treatment. The investigators expect that the combined treatment applied at the acute stage of PLP will have synergistic effects on PLP intensity and thus avert its chronification. In addition, it will reduce phantom sensations, and negative affect, and will improve the sense of body ownership and agency and endogenous inhibition efficiency.

Research design: This randomized-controlled double-blinded study will be held at Israel's 3 largest rehabilitation centers. The study consists of 3 randomized patient arms (36 in each): (1) no-intervention, natural-course group; (2) MT + sham tDCS; (3) MT + real tDCS.

MT and tDCS neuromodulatory interferences will be self-administered and consist of 20 sessions, completed during 4 weeks. The researchers outcome measures include: primary outcome: pain intensity, network-related behavioral markers, and amputation-related clinical characteristics. The data gathered will be collected at 5 timepoints.

Research novelty and innovation: The researchers proposed model will provide insights on the prevention of PLP and, potentially, other neurological pathologies involving the dysfunction of sensory systems and integration and body perception.

DETAILED DESCRIPTION:
Approximately 80% of amputees experience PLP, often severe, for years after amputation and most amputees will experience phantom limb sensations, including kinetic, proprioceptive (i.e. feeling of length or volume) and exteroceptive sensations (e.g. touch, pressure, itching). Treatment options for PLP have generally been limited, and there is no clear consensensus on the optimal treatment regimen. In PLP maladaptive plasticity associated with sensory defferentation following an amputation is one of the contributors for excessive pain.

This research project will focus on combined known neuromodulatory interventions of MT and tDCS, applied for the first time at the acute state of PLP in traumatic and non-traumatic amputees, with an aim to prevent maladaptive plasticity associated with PLP chronification and chronicity.

MT and tDCS related literature is based on data collected from patients who already developed PLP for years, before enrollment in the study. The investigators suggest that tDCS and MT applied at the acute stage of PLP will have synergistic effects on PLP intensity and thus avert its chronification. The researchers rationale is based on recent evidence from basic neuroscience on the phantom perception of other non-pain sensory modalities and the neuroscience of chronification of other pain conditions.

The fundamental mechanism for PLP suggests initial changes at the peripheral nervous system, including loss of afferent somatosensory input and exaggerated input from ectopic activity generated in the axotomized nociceptive neurons. Subsequent central changes include thalamic and cortical functional reorganization in the sensorimotor cortex, manifested as maladaptive cortical reorganization: an "invasion" of neighboring areas to the representation of the amputated limb.

Evidence in the literature suggests that the 2 noninvasive neuromodulation techniques- MT and tDCS applied to motor cortex (M1-tDCS)-may interfere with the maladaptive plasticity accompanied PLP and respectively will reduced PLP and negative affects. With MT, the moving, healthy limb reflected in the mirror makes the missing limb appear intact and functioning. The analgesic effect attributed to MT likely results from enhanced coherence between sensory feedback and motor command, counterbalancing the amputation-induced maladaptive neuroplasticity. In chronic PLP, MT conducted over several weeks reversed sensorimotor reorganization and reduced PLP intensity, suggesting a correlation between reorganization and PLP. MT also modulates the activity of the multisensory integration network to resolve the post-amputation perceptual incongruence, and modulates the activity of networks which help integrate the perceptual and motor areas to affect the sense of body ownership and agency. Indeed, an improved sense of agency has been reported after MT. Yet, these studies examined patients with chronic PLP and found mild analgesic effects. The investigators argue that MT applied at the acute PLP stage may interfere with the maladaptive plasticity of the multisensory integration network, and accordingly will improve the sense of agency and ownership over phantom limb, and reduce PLP intensity.

Motor areas (M1) stimulation through neuromodulation techniques alters the functional connectivity between brain areas, thus modulating brain networks rather than just affecting the local stimulation target. Specifically, it modulates ascending sensory input; brain areas of the fronto-striatal circuit, limbic brain areas, and midbrain nuclei involved in descending pain inhibition. Thus, tDCS applied to M1 may modulate brain areas composed of the subcircuits connected to mPFC and the salience network , i.e., areas presumably involved in pain chronification and chronicity. Although the electrical current only affects the cortex below the electrode, remote cortical and subcortical connected areas are affected as well. Previous work has described two putative analgesic effects of anodal M1 tDCS: 1) modulation of thalamic activity by descending corticothalamic pathways originating in the primary motor cortex and 2) inhibition of the primary somatosensory cortex via corticocortical pathways. Clinically, tDCS has immediate, sustained, and long-term analgesic effects. The investigators expect that M1-tDCS will restore the function of the mPFC and the salience network, and will thus improve endogenous pain inhibition, reduce PLP intensity and negative affect, yet will not eliminate pain chronification.

Because MT and tDCS, when given alone, produced only mild analgesic effects, their clinical adoption was limited. Soler et al. were the first to study the analgesic effects of a combination of visual illusion (similar to MT) and tDCS on neuropathic pain after spinal cord injury. The investigators found that the combination reduced pain intensity significantly more than did any single intervention; this effect lasted at least 12 weeks post-treatment. Gunduz et al. found no cumulative effect of MT and tDCS on patients with limb amputation. Whether studies examined the clinical effects of MT, tDCS, or a combination of both, the entire literature is based on data collected from patients with chronic PLP and did not consider time since amputation as an exclusion criterion. Therefore, time since amputation might be a key factor in the efficacy of these treatments. In patients who had only recently undergone amputation, the abnormal neuroplasticity might not yet be fixated; therefore, counterbalancing it should be easier. A preliminary study from Treister's lab is the first to show that a combination of MT and tDCS applied at the acute stage of PLP can prevent PLP chronification. Considering Treister's preliminary results and given that MT and M1-tDCS exert neuroplastic effects on different neural networks with similar outcome (i.e., PLP intensity), the investigators expect that a combination of MT and tDCS applied at the acute stage of PLP will have synergistic effects on PLP intensity and thus avert its chronification.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥18);
* Amputation of a single limb ≤12 weeks ago; during this period of time, 80% of amputees develop PLP. Both upper and lower limb amputees are included to increase feasibility;
* Acute PLP stage (2 weeks since first report), with intensity ≥3 on a 0-10 VAS;
* No change in medication in past week, excluding pro re nata analgesics;
* Can understand the study's purpose and instructions;
* Agrees to participate and to provide written informed consent.

Exclusion Criteria:

* Stump wound not healed;
* Other psychological, psychiatric, or neurological conditions;
* Contraindications for tDCS or magnetic resonance imaging (MRI) (MRI data will not be analyzed in the proposed PhD project), including previous seizure, loss of consciousness due to head injury, metal in the head, implanted devices, claustrophobia, a skin condition or an unhealed wound on the scalp, and possibility of being pregnant;
* Inability to provide informed consent or understand or carry out the experiment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
A 0-100 VAS of mean pain intensity during one week | Pain will be compared between baseline and 4 weeks after the end of the 4 weeks intervention (meaning, comparing baseline to timepoint number 3, which is exactly 8 weeks from the end of the baseline week)
  completed during 7 days, will be used to capture the weekly average of pain intensity (0 = no pain to 100 = the worst imaginable pain, via pain diary). This data will be used either in its raw, continuous form or as a transformed dichotomous variable, yes/no chronic PLP. A cutoff value of PLP intensity ≤20/100 will be used, because from a clinical perspective, pain intensity ≤20 is considered low and will seldom prompt a request for analgesic treatment.

SECONDARY OUTCOMES:
Sense of ownership and agency over phantom limb | Sense of ownership and agency over phantom limb will be compared between baseline and 4 weeks after the end of the 4 weeks intervention (meaning, comparing baseline to timepoint number 3, which is exactly 8 weeks from the end of the baseline week)
  Sense of ownership and agency over phantom limb will be a behavioral marker for function of the multisensory integration network. It will be evaluated using a self-report questionnaire with demonstrated sensitivity to detect changes after MT. Six of the questionnaire's 8 items (on a 5-point Likert scale) will be used to assess sense of ownership and agency of upper limb and will be adjusted for the lower limb. Mean scores of 3 questions will evaluate the sense of ownership, and 3 others, the sense of agency, as recommended.
The Hospital Anxiety and Depression Scale (HADS) | Anxiety and Depression will be compared between baseline and 4 weeks after the end of the 4 weeks intervention (meaning, comparing baseline to timepoint number 3, which is exactly 8 weeks from the end of the baseline week)
  The researchers' marker for function of the fronto-striatal-amygdala circuit, will be assessed via the Hospital Anxiety and Depression Scale (HADS), a self-report 14-item questionnaire focusing on nonphysical symptoms, which measures anxiety and depression, both demonstrated associations with changes in fronto-striatal connectivity. The HADS uses a 0-21 scoring scale, with each item rated on a 4-point Likert scale (0-3). A score of 0-7 is considered normal, 8-10 indicates a mild disorder, 11-14 suggests a moderate disorder, and 15-21 points to a severe disorder.
The Short Form McGill Pain Questionnaire | The Affective qualities of pain will be compared between baseline and 4 weeks after the end of the 4 weeks intervention (meaning, comparing baseline to timepoint number 3, which is exactly 8 weeks from the end of the baseline week)
  The researchers' marker for function of the fronto-striatal-amygdala circuit, will also be assessed via the Short Form McGill Pain Questionnaire, which assesses various affective qualities of pain and has demonstrated validity in neuropathic populations. Four affective descriptors rated on a 0-10 numerical rating scale will be summarized.
The Conditioned Pain Modulation (CPM) | The CPM score will be compared between baseline and 4 weeks after the end of the 4 weeks intervention (meaning, comparing baseline to timepoint number 3, which is exactly 8 weeks from the end of the baseline week)
  Endogenous pain inhibition will be a psychophysical marker for function of the fronto-PAG circuit. It will be evaluated by the conditioned pain modulation (CPM) paradigm, based on the systemic pain-inhibits-pain phenomenon. The conditioning stimulus will be administrated by immersing the palm in a cold-water bath (14°C). The test stimulus applied on the contralateral (to the conditioning stimulus) lower leg will include individually calibrated heat pain stimulus applied for 20 sec, while averaging pain intensity scores on a VAS Scale (0=no pain, 100= the worst imaginable pain) reported at time 0, 10, and 20 sec. CPM is calculated by subtracting pain scores of the test stimulus given alone from those given with the conditioning stimulus, as recommended.
Frequency of PLP paroxysms | Frequency of PLP paroxysms will be compared between baseline and 4 weeks after the end of the 4 weeks intervention (meaning, comparing baseline to timepoint number 3, which is exactly 8 weeks from the end of the baseline week)
  Frequency of PLP paroxysms, known to be correlated with PLP intensity or to be affected by neuromodulation techniques applied in PLP, will be evaluated daily for 1 week. Paroxysm will be defined as a period when PLP clearly increases above background pain level; frequency will be evaluated by the average value of the daily score on a 0-100 VAS (0="never during the day" to 100="very frequently").
Stump pain | Stump pain will be compared between baseline and 4 weeks after the end of the 4 weeks intervention (meaning, comparing baseline to timepoint number 3, which is exactly 8 weeks from the end of the baseline week)
  Stump pain, known to be correlated with PLP intensity or to be affected by neuromodulation techniques applied in PLP, will be evaluated daily for 1 week. It will be evaluated by the average value of the daily score on a 0-100 VAS (0="not painful at all" to 100="the worst imaginable pain").
Phantom sensations | Phantom sensations be compared between baseline and 4 weeks after the end of the 4 weeks intervention (meaning, comparing baseline to timepoint number 3, which is exactly 8 weeks from the end of the baseline week)
  Phantom sensations, known to be correlated with PLP intensity or to be affected by neuromodulation techniques applied in PLP, will be evaluated daily for 1 week. It will be evaluated by the average value of the daily score on a 0-100 VAS (0="no sensations" to 100="very intense").
Telescoping | Telescoping be compared between baseline and 4 weeks after the end of the 4 weeks intervention (meaning, comparing baseline to timepoint number 3, which is exactly 8 weeks from the end of the baseline week)
  Telescoping, known to be correlated with PLP intensity or to be affected by neuromodulation techniques applied in PLP, will be evaluated daily for 1 week. Telescoping will be evaluated by the average value of the daily score on a 0-100 VAS (0="no telescoping sensations" to 100="very intense telescoping sensations").

CONTACTS AND LOCATIONS:
Overall Officials: Roi Treister, PhD, Study Director — University of Haifa Faculty of Social Welfare and Health Sciences
Locations (3):
- Israel (3):
  - Loewenstein Hospital, Raanana, Israel
  - Reut Medical Center, Tel Aviv, Israel
  - Sheba Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: Yes